CLINICAL TRIAL: NCT07124091
Title: The Effect of a Micro-Appreciation Intervention (Three-Things Journal Application) on Caregiver Burden, Family Functioning, and Happiness Levels for Mothers of Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, MÜJDE KERKEZ, Assist. Prof. Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0000-0002-5515-2752
Record Dates: First submitted 2025-07-28; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Parental Stress
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomyzed control
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Event Writing Intervention Group (Experimental): Mothers in this group will be asked to write down three positive events each day for four weeks as part of a positive psychology journaling intervention.
  Interventions: Behavioral: Positive Event Writing Intervention
- Control Group (No Intervention): Mothers in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Positive Event Writing Intervention — Mothers in the intervention group will be asked to write down three positive events each day for four weeks as part of a positive psychology journaling activity..
  Arms: Positive Event Writing Intervention Group

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder in which individuals experience significant difficulties in social interaction, communication, and repetitive behaviors. Families of children with ASD, especially mothers, face a high level of physical, emotional, and psychological caregiving burden while trying to adapt to their children's developmental needs. Constant caregiving responsibilities increase the risk of burnout, stress, and depression in mothers, while also negatively impacting family functioning and life satisfaction. Mothers of children with ASD require greater emotional resilience, self-regulation, and social support than those in traditional parenting roles.

In this context, interventions that support psychological well-being offer important strategies that can help mothers cope with the burden of care. In recent years, positive psychology-based interventions have been shown to positively contribute to individuals' mental health and are effective in increasing subjective well-being. Positive psychology approaches help individuals recognize and focus on the positive aspects of their lives, reducing stress levels and increasing psychological resilience. One such approach, micro-appreciation interventions, aims to increase individuals' positive emotional experiences by consciously focusing on small but significant positive events they encounter in their daily lives. Micro-appreciation interventions change individuals' perceptual frameworks, encouraging them to focus on positive moments instead of negative experiences. Such interventions stand out as an effective method for reducing the psychological and physiological effects of stress, increasing positive emotions, and improving overall life satisfaction.

One micro-appreciation intervention, the "Three Things Journal," is a simple yet effective strategy that involves individuals writing down three positive events they appreciate in their lives each day. Research has shown that this practice is effective in increasing individuals' awareness of positive experiences, reducing levels of depression and anxiety, and increasing subjective well-being. Regularly experiencing positive emotions strengthens individuals' ability to cope with challenges and increases their psychological resilience and optimism. Especially for individuals under intense stress, such small but regular practices can yield greater psychological benefits in the long term.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Willing to participate in the study
* Able to read and understand Turkish
* Being a mother of a child with special needs

Exclusion Criteria:

* Younger than 18 years
* Unwilling to participate in the study
* Unable to read or understand Turkish
* Not having a child with special needs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Happiness Levels as Measured by the Oxford Happiness Questionnaire - Short Form (OHQ-SF) | Baseline and Week 5
  The Oxford Happiness Questionnaire - Short Form (OHQ-SF) is a 7-item scale used to assess individual levels of happiness. Each item is rated on a Likert scale. Total scores range from 0 to 28, with higher scores indicating greater happiness. The Turkish adaptation was validated by Doğan and Çötok (2011) with a reliability coefficient (Cronbach's alpha) of .74 and test-retest reliability of .85.
Change in Caregiver Burden as Measured by the Zarit Burden Interview (ZBI) | Baseline and Week 5
  The Zarit Burden Interview (ZBI) is a 22-item self-report instrument assessing perceived burden among caregivers. Each item is scored from 0 ("Never") to 4 ("Nearly Always") using a 5-point Likert scale. The total score ranges from 0 to 88, with higher scores indicating greater caregiver burden. The Turkish version was validated by İnci and Erdem (2007), with a Cronbach's alpha of .90.
Change in Family Functioning as Measured by the Family APGAR Scale | Baseline and Week 5
  The Family APGAR Scale is a 5-item measure of satisfaction with family functioning across five dimensions: adaptability, partnership, growth, affection, and resolve. Each item is rated on a 3-point scale from 0 ("Rarely") to 2 ("Almost always"). Total scores range from 0 to 10, with higher scores indicating greater satisfaction with family functioning. Scores between 0-3 suggest low satisfaction, 4-6 moderate satisfaction, and 7-10 high satisfaction. The Turkish version was validated by Özcan et al. (2011), with a Cronbach's alpha of .793.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman University, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In this study, the names of the studies will be shared in accordance with the rules of the Declaration of Helsinki and the study results will be presented with analyses.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT07124091/ICF_000.pdf